CLINICAL TRIAL: NCT06987136
Title: A Randomized Clinical Trial Comparing Transversus Thoracic Muscle Plane Block, Erector Spinae Plane Block and Paravertebral Block for Analgesia in Patients Undergoing Video-Assisted Thoracic Surgery
Brief Title: Transversus Thoracic Muscle Plane Block, Erector Spinae Plane Block and Paravertebral Block for Analgesia in Video-Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdalsattar Elmohasseb, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1184/4/25.
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Transversus Thoracic Muscle Plane Block; Erector Spinae Plane Block; Paravertebral Block; Analgesia; Video-Assisted Thoracic Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transversus thoracic muscle plane block group (Experimental): Patients will receive a transversus thoracic muscle plane block.
  Interventions: Other: Transversus thoracic muscle plane block
- Erector spinae plane block group (Experimental): Patients will receive an erector spinae plane block.
  Interventions: Other: Erector spinae plane block
- Thoracic paravertebral block group (Experimental): Patients will receive a thoracic paravertebral block.
  Interventions: Other: Thoracic paravertebral block

INTERVENTIONS:
Other: Transversus thoracic muscle plane block — Patients will receive a transversus thoracic muscle plane block.
  Arms: Transversus thoracic muscle plane block group
Other: Erector spinae plane block — Patients will receive an erector spinae plane block.
  Arms: Erector spinae plane block group
Other: Thoracic paravertebral block — Patients will receive a thoracic paravertebral block.
  Arms: Thoracic paravertebral block group

SUMMARY:
The aim of this study is to compare the transversus thoracic muscle plane block (TTPB), erector spinae plane block (ESPB), and thoracic paravertebral block (TPVB) for postoperative analgesia in patients undergoing video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
Traditionally, resection is done via a thoracotomy. Still, video-assisted thoracoscopic surgery (VATS) provides significant advantages over open thoracotomy procedures, including reduced surgical pain, improved postoperative pulmonary function, reduced mortality, shortened hospital stay. It has emerged as a minimally invasive alternative.

Thoracic paravertebral block (TPVB) is a regional anesthetic technique in which local anesthetic (LA) is administered inside the thoracic paravertebral space (TPVS), which contains the intercostal spinal nerves, spinal dorsal rami, rami communicants, sympathetic chain, intercostal vessels, and fatty tissue.

The erector spinae plane block (ESPB) is an interfascial regional anesthesia block for thoracic analgesia which can be performed by superficial or deep needle approach.

Transversus thoracic muscle plane block (TTPB) is a newly developed technique in which LA is injected into the fascial plane between the transversus thoracic muscle and the internal intercostal muscles for blocking the anterior cutaneous branches of intercostal nerves from thoracic (Th) 2 to Th 6.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for video-assisted thoracic surgery under general anesthesia.

Exclusion Criteria:

* Body mass index >30 kg/m2.
* Coagulopathy.
* History of opiate abuse.
* Pre-existing chronic pain.
* Allergy to local anesthetics or analgesics.
* Infection at the site of injection.
* Mental or neurological disorders.
* Operation converted to open thoracotomy.
* Renal dysfunction (glomerular filtration rate (GFR) < 50 ml/min).
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-24 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the Visual Analogue Scale (VAS) > 3 to be repeated after 30 min if pain persists until the VAS < 4.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively, before the block is performed, and every 15 minutes until the end of surgery.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively, before the block is performed, and every 15 minutes until the end of the surgery.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as pneumothorax, bradycardia, hypotension, nausea, vomiting, pruritis, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.